CLINICAL TRIAL: NCT05061498
Title: Impact of Pacing Output and Cycle Length on QRS Morphology in Ablation of Premature Ventricular Contractions
Brief Title: Impact of Pacing Output and Cycle Length on QRS Morphology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pacemap-Study
Record Dates: First submitted 2021-05-11; First posted 2021-09-29 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: PVC - Premature Ventricular Complex; Catheter Ablation
Keywords: Catheter ablation of PVC; Pacemapping
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional Pacing maneuvers (Other): In all study participants additional pacing maneuvers (cycle lenght and output) are performed
  Interventions: Diagnostic Test: Additional Pacing maneuvers

INTERVENTIONS:
Diagnostic Test: Additional Pacing maneuvers — In order to determine the optimal setting for pacemapping in all participants additional pacing maneuvers (output and cycle length) are performed

SUMMARY:
Current recommendations for pacemapping are based on expert opinion and animals models. Present study sought to evaluate the influence of different parameters of pacemapping on QRS morphology. Pacemapping is performed with different cycle length (fixed burst vs. coupling interval) and stimulation output (maximum output vs. threshold) and resulting QRS complexes are compared to clinical PVC and the standard of care to determine the optimal parameter setting in pacemapping.

DETAILED DESCRIPTION:
Pacemapping is a common technique to determine to origin of ventricular ectopy during catheter ablation of premature ventricular contractions (PVC). During the pacemapping process an electrical pacing stimulus is applied via the ablation catheter and the resulting QRS complex is compared the clinical target PVC. The higher the consistency between the stimulated QRS complex and the clinical PVC, the nearer the catheter is located to the origin of ectopy.

Current recommendations for the execution of pacemapping are based on expert opinion and animals models. The investigators sought to assess for the first time in a clinical real life setting the different parameters for pacemapping (i.e. Cycle length and stimulation output). Therefore during the pacemapping process in routine PVC ablation pacing is performed with different cycle length (fixed burst vs. coupling interval of PVC) and different electrical output (maximum output vs. stimulation threshold). The resulting QRS morphologies are on the one hand compared to the ablation target (clinical PVC) and on the other hand to the suggest standard of care (Coupling interval at pacing threshold) to determine the optimal setting of parameters in pacemapping.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing PVC ablation

Exclusion Criteria:

* patients <18 years
* patients not able to consent
* pregnancy
* contraindication for PVC ablation
* unavailability of vascular access
* patients with complex congenital heart disease
* expected hemodynamical instability during pacemapping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Template Matching with clinical PVC | Immediately during PVC ablation. No follow up intended.
  Different pacing settings are applied in order to determine the optimal Consistency between paced QRS complex and clinical PVC

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Lüker, MD, Principal Investigator — Heart Center University of Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No